CLINICAL TRIAL: NCT01750606
Title: An MRI Investigation of Soft Tissues in Total Hip Arthroplasty
Acronym: MoM_MRI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GH04; PS110005-28 (Other: FDA)
Record Dates: First submitted 2012-11-06; First posted 2012-12-17 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-07

CONDITIONS: Tissue Reaction; Elevated Blood Ion Levels

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (6):
- pre-THA: Patients who are planned but have not yet received a total hip arthroplasty. No intervention or treatment - blood draw only to be used as a surrogate baseline for metal ion exposure.
- Metal-on-Poly: Patients receiving a Biomet metal on poly hip implanted between January 1, 2003 and December 31, 2006.
- M2a Magnum hip: Patients receiving a Biomet M2a Magnum hip implanted between January 1, 2006 and January 1, 2011.
- M2a38 hip: Patients receiving a Biomet metal on metal M2a38 hip implanted between January 1, 2004 and December 31, 2006.
- M2a Ringloc hip: Patients receiving a Biomet M2a Ringloc metal on metal hip implanted between January 1, 2002 and December 31, 2004.
- M2a Taperloc hip: Patients receiving a Biomet M2a Taperloc metal on metal hip implanted between January 1, 2002 and December 31, 2003.

SUMMARY:
Retrospective study to comply with FDA's post-market surveillance order. The purpose of the study is to contact patients who have received a Biomet metal-on-metal product as their primary total hip arthroplasty device. Patients who have not been revised prior to contact will be asked to submit to a blood draw, clinical exam and MRI.

DETAILED DESCRIPTION:
This study has been designed to estimate the prevalence of soft tissue changes following primary THA surgery in patients having received one of five Biomet implant types; a MOP primary THA, an M2a 38, M2a Taper, M2a Ringloc and M2a Magnum MOM primary THA device in 308-436 total patients at four centers.

The primary objective of the study is to estimate the prevalence of soft tissue changes in unbiased MoM and MoP samples. Secondary objectives are to evaluate whether the occurrence of soft tissue changes is related to any of several potential covariates including patient and implant characteristics and time in situ.

ELIGIBILITY:
Inclusion Criteria:

* patient meets the sampling plan requirements

Exclusion Criteria:

* patient is contraindicated for MRI
* patient fails to consent for the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received the indicated implants at one of four participating centers and who meet the sampling plan requirements.
Sampling Method: Non-Probability Sample
Enrollment: 436 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of symptomatic and asymptomatic Metal-on-Metal and Metal-on-Poly patients (via a proportion) with a soft tissue mass | patients 3 years post-implantation up to 6 years post implantation
  Compare the proportion of symptomatic and asymptomatic Metal-on-Metal patients with a soft tissue mass to the proportion of Metal-on-Poly patients with soft tissue masses.

SECONDARY OUTCOMES:
Metal ion concentrations in whole blood and serum | 1-10 year post implantation, depending on cohort
  Determine metal ion concentrations in whole blood and serum and assess whether findings correlate to any other variable such as pain, implant type, time since surgery and presence of ALTR.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schenck, Ph.D., Study Director — Zimmer Biomet
Locations (5):
- United States (5):
  - Ortho Michigan, Flint, Michigan
  - Joint Implant Surgeons, New Albany, Ohio
  - Midlands Orthopaedics, Columbia, South Carolina
  - Texas Center for Joint Replacement, Plano, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided